CLINICAL TRIAL: NCT02708693
Title: Efficacy of Combined Ultrasound Guided Steroid Injection and Splinting in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-05-021A
Record Dates: First submitted 2016-01-05; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2013-04

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Triamcinolone Acetonide; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental: steroid injection and splinting (Experimental): ultrasound-guided steroid injection using 1ml of 10 mg (10mg/ml) triamcinolone acetonide (Shincort) mixed with 1 ml of 2% lidocaine hydrochloride (Xylocaine) and a customized volar thermoplastic wrist splint
  Interventions: Drug: Triamcinolone Acetonide; Device: thermoplastic wrist splint; Drug: lidocaine hydrochloride
- steroid injection (Active Comparator): ultrasound-guided steroid injection using 1ml of 10 mg (10mg/ml) triamcinolone acetonide (Shincort) mixed with 1 ml of 2% lidocaine hydrochloride (Xylocaine)
  Interventions: Drug: Triamcinolone Acetonide; Drug: lidocaine hydrochloride

INTERVENTIONS:
Drug: Triamcinolone Acetonide — ultrasound-guided injection using 1ml of 10 mg (10mg/ml) triamcinolone acetonide (Shincort)
  Other Names: triamcinolone acetonide 10mg/ml (shincort, YSP, Taiwan)
Device: thermoplastic wrist splint — thermoplastic wrist splint with wrist placed in a neutral position
  Arms: experimental: steroid injection and splinting
Drug: lidocaine hydrochloride — ultrasound-guided injection using 1 ml of 2% lidocaine hydrochloride (Xylocaine)
  Other Names: lidocaine hydrochloride (Xylocaine)

SUMMARY:
To compare the effectiveness of ultrasound guided-steroid injection plus splinting to that of steroid injection alone using clinical and electrophysiological parameters in patients with carpal tunnel syndrome

DETAILED DESCRIPTION:
This is a prospective, single-blinded randomized controlled study. Patient with CTS were randomly assigned to group receiving ultrasound guided steroid injection and group receiving ultrasound guided corticosteroid injection and splinting. The steroid injection was using 1ml of 10 mg (10mg/ml) triamcinolone acetonide (Shincort) mixed with 1 ml of 2% lidocaine hydrochloride (Xylocaine). The inclusion criteria included an age of more than 18 years and typical signs of CTS according to American Academy of Neurology criteria lasting for at least 3 months. The diagnosis of CTS was confirmed by electrophysiological tests.The exclusion criteria included the following: presence of thenar atrophy; existence of disorders such as hypothyroidism, diabetes mellitus, chronic renal failure, or rheumatoid arthritis; any accompanying orthopedic or neurologic disorders that could mimic CTS such as cervical radiculopathy, polyneuropathy, proximal median nerve entrapment, or thoracic outlet syndrome; prior steroid injection into the affected carpal tunnel or carpal tunnel surgery; history of distal radius fracture; pregnancy or lactation; regular use of systemic NSAIDs or corticosteroids; and known allergy to corticosteroids and local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of CTS
2. The diagnosis of CTS was confirmed by electrophysiological tests.

Exclusion Criteria:

1. presence of thenar atrophy
2. existence of disorders such as hypothyroidism, diabetes mellitus, chronic renal failure, or rheumatoid arthritis; any accompanying orthopedic or neurologic disorders that could mimic CTS such as cervical radiculopathy, polyneuropathy, proximal median nerve entrapment, or thoracic outlet syndrome
3. prior steroid injection into the affected carpal tunnel or carpal tunnel surgery
4. history of distal radius fracture
5. pregnancy or lactation
6. regular use of systemic NSAIDs or corticosteroids
7. known allergy to corticosteroids and local anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the scores on the Boston Carpal Tunnel Questionnaire (BQ). | at 2, 6, 12 weeks
  The BQ was interviewed-administered to assess the severity of symptoms and functional status.

SECONDARY OUTCOMES:
Change from Baseline in Median nerve distal motor latency | at 2, 6, 12 weeks
  or the motor studies, the CMAPs were obtained via surface electrodes placed on the abductor pollicis brevis muscle. The active recording electrode was placed on the muscle belly, and the reference electrode was placed on the tendon insertion. The median nerve was stimulated 8 cm proximal to the active recording electrode. Distal motor latencies were measured from the onset of stimulus artifact to the onset of the CMAP
Change from Baseline in sensory nerve conduction velocity | at 2, 6, 12 weeks
  SNAPs were obtained using an antidromic method and recorded by surface electrodes placed at the proximal and distal interphalangeal joints of the index finger for the median nerve and the same joints of the little finger for the ulnar nerve. The median nerves were stimulated at the wrist at a distance of 14 cm from the wrist to the active electrode. Distal sensory latencies were measured from the onset of the stimulus artifact to the onset of the SNAP. SNCV was calculated dividing the distance of 14 cm by the distal sensory latency.
Change from Baseline in compound muscle action potential amplitude (CMAP) | at 2, 6, 12 weeks
  the CMAPs were obtained via surface electrodes placed on the abductor pollicis brevis muscle. The active recording electrode was placed on the muscle belly, and the reference electrode was placed on the tendon insertion. The median nerve was stimulated 8 cm proximal to the active recording electrode. The amplitude of CMAP were measured from baseline to negative peak.
Change from Baseline in sensory nerve action potential amplitudes. | at 2, 6, 12 weeks
  SNAPs were obtained using an antidromic method and recorded by surface electrodes placed at the proximal and distal interphalangeal joints of the index finger for the median nerve and the same joints of the little finger for the ulnar nerve. The median nerves were stimulated at the wrist at a distance of 14 cm from the wrist to the active electrode. The amplitude of SNAP were measured from baseline to negative peak.
Change from Baseline in self-reported pain intensity | at 2, 6, 12 weeks
  Patients were asked to indicate the intensity of their average level of pain for the wrist-hand region within the past 1 week, using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable).
change from Baseline in Cross sectional area | at 2, 6, 12 weeks
  The CSA of the median nerve was measured using ultrasound at 2 levels: at the carpal tunnel inlet (CSA-I; immediately prior to the proximal margin of the flexor retinaculum) and in the mid-carpal tunnel (CSA-M; at the level of the pisiform bone and scaphoid tubercle). The CSA within the surrounding hyperechoic rim was measured. The CSA was measured using a continuous boundary trace of the nerve and was directly calculated using the area measurement software included with the ultrasonography device
change from Baseline in flattening ratio | at 2, 6, 12 weeks
  The flattening ratio was measured only at the mid-tunnel (FR-M) using ultrasound. FR was calculated by dividing the horizontal diameter of the nerve by the vertical diameter.